CLINICAL TRIAL: NCT02736669
Title: Fixed Versus Variable Energy Reduction During Behavioral Obesity Treatment
Brief Title: CARE Trial: Comparing Different Levels of Calorie Reduction for Weight Loss
Acronym: CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Gareth R. Dutton PhD, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-150303008; R01DK103863 (NIH)
Record Dates: First submitted 2016-04-04; First posted 2016-04-13 (Estimated); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Overweight; Obesity
Keywords: weight loss; body weight; behavioral
MeSH Terms: conditions — Overweight; Obesity; Weight Loss; Body Weight; Behavior

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fixed Energy (or Calorie) Reduction (Active Comparator): Participants randomly assigned to this arm will be instructed to reduce their food intake by a moderate amount and stay at this level of moderate reduction until their weight loss goal is achieved.
  Interventions: Behavioral: Energy Reduction
- Variable Energy (or Calorie) Reduction (Experimental): Participants randomly assigned to this arm will be instructed to alternate between two levels of calorie reduction. One level will be a small amount of calorie reduction, while the other will be a more significant amount of calorie reduction. At the instruction of the research team, participants will periodically alternate back and forth between these two goals until their weight loss goal is achieved.
  Interventions: Behavioral: Energy Reduction

INTERVENTIONS:
Behavioral: Energy Reduction

SUMMARY:
This research study will compare two weight loss programs that provide different recommendations for how to reduce your energy (or calorie) intake to achieve weight loss in an effort to determine if fixed calorie reduction or varied calorie reduction is more effective for weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-75
* Body mass index (BMI) 30-50 kg/m2

Exclusion Criteria:

* Uncontrolled hypertension (blood pressure >160/100 mm Hg)
* Any of the following other medical conditions: myocardial infarction or cerebrovascular accident within the last six months; unstable angina within the past six months; congestive heart failure; cancer requiring treatment in past five years (exception: non-melanoma skin cancer); serious infectious diseases (e.g., self-reported HIV); chronic hepatitis; cirrhosis; chronic malabsorption syndrome; chronic pancreatitis; chronic lung diseases or orthopedic problems that limit physical activity
* Current use of any of the following medications: antipsychotic agents, monoamine oxidase inhibitors, systemic corticosteroids, antibiotics for HIV or TB, or chemotherapeutic drugs; prescription weight loss medications (past six months)
* Unwilling or unable to do any of the following: give informed consent; read English at the 5th grade level; accept random assignment; travel to the intervention site
* Likely to relocate out of the area in the next 2 years
* Participation in another randomized research project
* Weight loss > 10 pounds in past six months
* History of bariatric surgery
* Major depressive or psychiatric disorder, or excessive alcohol intake
* Potential participants living farther than 30 miles driving distance from UAB will be excluded from the study.
* Potential participants (female) that are pregnant or plan to become pregnant in the next 18 months will be excluded from participation in the study. This is a weight loss study and weight gain/loss due to pregnancy and/or delivery would confound study results. Additionally, weight loss is not recommended for pregnant women.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Measure change in body weight (kg) from baseline to follow-up assessments | Baseline, 6 months, 18 months
  Participants will be weighed by body scale in kilograms

SECONDARY OUTCOMES:
Resting energy expenditure | 6, 12, and 18 months
  An indirect calorimeter with the ventilated hood technique will be used for the 30-minute measurement (the first 10 minutes will be excluded from analysis). The respiratory quotient will be calculated as the ratio of carbon dioxide production to oxygen consumption. Resting metabolic rate will be calculated from VO2 and VCO2 measurements using the Weir equation.
Body composition | 6, 12, and 18 months
  Assessed by full body DXA scan to evaluate percentage of body fat.
Laboratory analyses | 6, 12, and 18 months
  Glucose, lipids, and insulin will be analyzed using blood samples.
Blood pressure | 6, 12, and 18 months
  After a 5 minute seated rest, three measurements using an automated blood pressure device will be taken to obtain the average systolic and diastolic blood pressures.
Hormones - ghrelin | 6, 12, and 18 months
  Total ghrelin will be assessed using blood samples.
Hormones - leptin | 6, 12, and 18 months
  Total leptin will be assessed using blood samples.
Satiety/hunger | 6, 12, and 18 months
  Visual analogue scales (VAS) will be used to measure subjective ratings of appetite. Participants will be asked to provide a rating in response to several questions (e.g., "How hungry did you feel this week? How much did you think about food this week?") using a 100-mm line ranging from "not at all" to "extremely".
Physical activity - objective | 6, 12, and 18 months
  Will be assessed via accelerometers worn by participants for seven days. Participants will be instructed to position the accelerometer at the right hip and to wear the device throughout the day except when sleeping, bathing, or participating in swimming or other water activities. These data will be used to estimate total minutes of moderate- to vigorous-intensity PA.
Physical activity - self-report | 6, 12, and 18 months
  Self-reported PA will also be assessed with the Paffenbarger Physical Activity Questionnaire (PPAQ). Both methods of PA measurement are included, as accelerometers provide objective information about total levels of activity, while the PPAQ provides additional details about the type and schedule of activities.
Treatment adherence | 6, 12, and 18 months
  Treatment adherence will be assessed by the number of treatment sessions attended as well as the number of self-monitoring forms completed, which have both been used as indicators of adherence in our previous work
Treatment novelty | 6, 12, and 18 months
  This construct will be evaluated with a 6-item measure of treatment reinforcement that assesses the extent to which participants enjoy and become less habituated to the behavioral strategies required for weight loss.
Treatment burden | 6, 12, and 18 months
  Behavioral burden of treatment will be assessed with a modified version of the Treatment Burden Questionnaire (TBQ), which includes 15 items measuring the burden of treatment, including behaviors of self-monitoring, dietary changes, maintaining physical activity, and the impact of treatment on social relationships.
Treatment satisfaction | 6, 12, and 18 months
  Participants will complete a modified version of the Treatment Satisfaction Questionnaire for Medication (TSQM) to assess attitudes and satisfaction regarding the weight loss intervention, energy prescriptions provided, and weight loss achieved. A composite score of treatment satisfaction will be calculated based on participants' responses.

CONTACTS AND LOCATIONS:
Overall Officials: Gareth R Dutton, PhD, Principal Investigator — University of Alabama at Birmingham, Department of Medicine, Division of Preventive Medicine
Locations (1):
- University of Alabama at Birmingham, Medical Towers Building, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
The PI will ensure all publications that result from project-related data will comply with the NIH public access policy and develop a system by which study data may be shared with other investigators within the scientific community. With UAB IRB permission, PI may develop a de-identified database, codebook, and mechanism by which data can be shared with qualified individuals/organizations. PI will keep a record of all individuals/res. teams who request/receive a copy of the data. Interested investigators will be asked to complete a request form stating specific aims of the analyses, analytic plan, available resources, proposed timeline, and goals. PI and team will review these requests to determine whether proposed analyses constitute significant exploration of the data, team has resources to complete request, and data will be adequately protected and managed. If any issues are problematic, PI and team will attempt to negotiate a fair resolution with investigators and NIH staff.